CLINICAL TRIAL: NCT04398368
Title: GEMINI: An Open-Label, Single-Arm, Phase II Study of Intraoperative Gemcitabine Intravesical Instillation in Patients Undergoing Radical Nephroureterectomy for Upper Tract Urothelial Carcinoma
Brief Title: Gemcitabine for the Prevention of Intravesical Recurrence of Urothelial Cancer in Patients With Upper Urinary Tract Urothelial Cancer Undergoing Radical Nephroureterectomy, GEMINI Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Focus research efforts on other projects.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen A. Boorjian, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-009444; NCI-2020-03336 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-009444 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2020-05-16; First posted 2020-05-21 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Stage 0a Renal Pelvis and Ureter Cancer AJCC v8; Stage 0a Renal Pelvis Cancer AJCC v8; Stage 0a Ureter Cancer AJCC v8; Stage 0is Renal Pelvis and Ureter Cancer AJCC v8; Stage 0is Renal Pelvis Cancer AJCC v8; Stage 0is Ureter Cancer AJCC v8; Stage I Renal Pelvis and Ureter Cancer AJCC v8; Stage I Renal Pelvis Cancer AJCC v8; Stage I Ureter Cancer AJCC v8; Stage II Renal Pelvis and Ureter Cancer AJCC v8; Stage II Renal Pelvis Cancer AJCC v8; Stage II Ureter Cancer AJCC v8; Stage III Renal Pelvis and Ureter Cancer AJCC v8; Stage III Renal Pelvis Cancer AJCC v8; Stage III Ureter Cancer AJCC v8; Stage IV Renal Pelvis and Ureter Cancer AJCC v8; Stage IV Renal Pelvis Cancer AJCC v8; Stage IV Ureter Cancer AJCC v8
MeSH Terms: conditions — Ureteral Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (gemcitabine hydrochloride) (Experimental): Patients receive gemcitabine hydrochloride intravesically for at least 1 hour at the time of RNU.
  Interventions: Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — Given intravesically
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011

SUMMARY:
This phase II trial studies how well gemcitabine works in preventing urothelial cancer from coming back within the bladder (intravesical recurrence) in patients with upper urinary tract urothelial cancer undergoing radical nephroureterectomy. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Instilling gemcitabine into the bladder during surgery, may reduce the chance of recurrence of upper urinary tract urothelial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of a single intraoperative intravesical instillation of gemcitabine hydrochloride (gemcitabine) at time of radical nephroureterectomy (RNU) for clinically localized upper tract urothelial carcinoma (UTUC) in preventing intravesical recurrence of urothelial cancer (UC) at one year.

SECONDARY OBJECTIVES:

I. To assess time to recurrence for entire duration of follow-up. II. To assess the qualitative and quantitative toxicities.

EXPLORATORY OBJECTIVES:

I. To stratify intravesical UC recurrence free survival by tumor grade, neoadjuvant chemotherapy, tumor stage, ureteral tumor location, and history of bladder cancer.

II. To assess incidence and time to development of muscle-invasive bladder cancer (MIBC).

OUTLINE:

Patients receive gemcitabine hydrochloride intravesically for at least 1 hour at the time of RNU.

After completion of study, patients are followed up at 2 weeks, and 3, 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of localized (clinical American Joint Committee on Cancer [AJCC] stage Ta-T4N0M0) low- and high-grade UC of the renal pelvis and/or ureter
* Plan to undergo RNU
* Creatinine < 2.2 mg/dL (194 mmol/L)
* Hemoglobin > 9 g/dL
* White blood cell count >= 3000/uL
* Platelet count > 75,000/uL and < 500,000/uL
* Serum bilirubin levels below 2 times the institution's upper limits of normal
* Alkaline phosphatase levels below 2 times the institution's upper limits of normal
* Aspartate aminotransferase levels below 2 times the institution's upper limits of normal
* Alanine aminotransferase levels below 2 times the institution's upper limits of normal
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 - 2
* Suitable candidate for surgery at the discretion of the investigator
* Patient must be capable of giving appropriate approved informed consent or have an appropriate representative available to do
* Patient with a prior malignancy allowed if adequately treated > 3 years ago with no current evidence of disease
* Women of childbearing potential (WOCBP) must have a negative pregnancy urine test within 28 days of registration, and be using an adequate method of contraception to avoid pregnancy prior to and for at least 6 months after gemcitabine instillation to minimize the risk of pregnancy
* Male patient who has a partner that is a WOCBP must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) and should avoid conceiving children prior to and for 6 months following gemcitabine instillation

Exclusion Criteria:

* Pure non-urothelial histology; urothelial carcinoma with differentiation allowed
* Evidence of nodal or distant metastases; enlarged retroperitoneal lymph nodes > 2 cm or histologically positive lymph nodes
* History of UC of the bladder within 12 months preceding RNU, or receipt of intravesical therapy within 6 months
* History of or current prostatic urethral, urethral, or contralateral upper tract UC
* Planned radical cystectomy at time of RNU
* Symptomatic urinary tract infection of bacterial cystitis (once satisfactorily treated, patients can enter the study)
* Patient with any current malignancy except for basal or squamous cell skin cancers, noninvasive cancer of the cervix, or any other cancer deemed to be of low-risk for progression or patient morbidity during the trial period (i.e. Gleason 6 prostate cancer, renal mass < 3 cm)
* Women who are pregnant or breastfeeding
* Prisoners or subjects who are involuntarily incarcerated
* Inability for adequate follow-up, including concerns for patient compliance or geographic proximity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Boorjian, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevention (Gemcitabine Hydrochloride)
Started | 25
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Prevention (Gemcitabine Hydrochloride)
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.38 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Urothelial Carcinoma Relapse-free Survival
Description: Number of participants without recurrence of Urothelial Carcinoma. Relapse-free survival will be assessed by cystoscopy and urine cytology.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Gemcitabine Hydrochloride)
Number analyzed (Participants) | 23
Participants | 14

2. Secondary Outcome: Time to Recurrence
Description: Number of days from Radical Nephroureterectomy to date of histologic proof of recurrence/relapse of Urothelial Carcinoma
Time Frame: Up to 1 year
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Prevention (Gemcitabine Hydrochloride)
Number analyzed (Participants) | 23
Days | 178.75 (136.39)

3. Secondary Outcome: Incidence of Adverse Events
Description: Adverse events will be categorized by grade and further distinguished as serious adverse events. Furthermore, they will be designated by each site as not related, unlikely, possible, probably, and definitely related to treatment adverse events. they will also be summarized and organized by organ system, with the number and percent of patients experiencing the adverse event at least once and the number of patients exposed. Adverse events will be described and analyzed qualitatively. Adverse events will be grouped into categories and numerically described.
Time Frame: Up to 2 years
Measure: Number; unit: Adverse Events
Arm/Group | Prevention (Gemcitabine Hydrochloride)
Number analyzed (Participants) | 23
Adverse Events | 213

4. Other Pre Specified Outcome: Incidence of Muscle-invasive Bladder Cancer
Description: Number of subject to experience muscle-invasive bladder cancer. Assessed by Urothelial Carcinoma on final pathology of Transurethral Resection of Bladder Tumor specimen or Urothelial Carcinoma on final pathology of radical cystectomy specimen.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Gemcitabine Hydrochloride)
Number analyzed (Participants) | 23
Participants | 4

5. Other Pre Specified Outcome: Time to Development of Muscle-invasive Bladder Cancer
Description: Defined as the time (days) from date of Radical Nephroureterectomy to date of histologic proof of Urothelial Carcinoma
Time Frame: Up to 2 years
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Prevention (Gemcitabine Hydrochloride)
Number analyzed (Participants) | 23
Days | 178.75 (136.39)

6. Other Pre Specified Outcome: Time to Death
Description: Defined as the time (days) from date of Radical Nephroureterectomy to date of death
Time Frame: Up to 2 years
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Prevention (Gemcitabine Hydrochloride)
Number analyzed (Participants) | 23
Days | 543 (379.97)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 24 months on all participants.
Arm/Group | Prevention (Gemcitabine Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 3/25
Serious Adverse Events (participants affected / at risk) | 4/25
Other Adverse Events (participants affected / at risk) | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevention (Gemcitabine Hydrochloride) (N=25)
atrioventricular block (complete) (Cardiac disorders) | 1 (1)
Cancer recurrence (Renal and urinary disorders) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nectrotic segment of small intestine (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevention (Gemcitabine Hydrochloride) (N=25)
abdominal pain (Gastrointestinal disorders) | 3 (3)
Hemmorrhage (Blood and lymphatic system disorders) | 2 (2)
Hematuria (Blood and lymphatic system disorders) | 3 (7)
Hearing Impared (Ear and labyrinth disorders) | 1 (1)
Sore Throat (General disorders) | 2 (3)
Facial Flushing (General disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (9)
Vomiting (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (4)
Nocturia (Renal and urinary disorders) | 4 (6)
Urinary Tract Infection (Infections and infestations) | 5 (8)
Hot Flashes (Nervous system disorders) | 2 (2)
Flank Pain (General disorders) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Penile Pain (General disorders) | 1 (1)
Scrotal Infection (Infections and infestations) | 1 (1)
Perineal pain (General disorders) | 1 (1)
Bladder Pain (Renal and urinary disorders) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1)
Testicular Pain (Reproductive system and breast disorders) | 3 (3)
Phantom Pain (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Chronic Kidney Disease (Renal and urinary disorders) | 4 (5)
Leg Edema (Vascular disorders) | 2 (2)
Fever (Immune system disorders) | 2 (2)
Loss of Appetite (Metabolism and nutrition disorders) | 1 (1)
Lightheadedness (Nervous system disorders) | 2 (2)
Weakness/Fatigue (Nervous system disorders) | 7 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Metallic taste (General disorders) | 1 (1)
Bladder Leak (Renal and urinary disorders) | 1 (1)
Hyperkalemia (Renal and urinary disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 2 (5)
Insomnia (Nervous system disorders) | 2 (2)
Scalp pain (General disorders) | 1 (1)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
Hypertension (General disorders) | 5 (6)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Scrotal Bruising (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Penile cancer (Reproductive system and breast disorders) | 1 (1)
Gross hematuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (3)
Abnormal liver function lab values (Hepatobiliary disorders) | 1 (1)
Anxiety (General disorders) | 1 (1)
Low platelet count (Blood and lymphatic system disorders) | 4 (7)
Elevated creatinine (Blood and lymphatic system disorders) | 5 (8)
Headaches (General disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Increased urinary frequency (Renal and urinary disorders) | 1 (1)
Hypotension (Nervous system disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Thoracic aorta calcification (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased vision function, unilateral (Eye disorders) | 1 (1)
Dry eye syndrome, bilateral (Eye disorders) | 1 (1)
Bladder Spasm (Renal and urinary disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Subcutaneous emphysema (General disorders) | 1 (1)
Hyperlipidemia (Blood and lymphatic system disorders) | 1 (1)
Fall (loss of balance) (General disorders) | 1 (1)
Pneumoperitoneum (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Weight loss (Metabolism and nutrition disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Elevated white blood call count (Blood and lymphatic system disorders) | 3 (3)
Unable to pass gas (Gastrointestinal disorders) | 1 (1)
Fissure, foot (Musculoskeletal and connective tissue disorders) | 1 (1)
Polyp, colon (Gastrointestinal disorders) | 2 (3)
Vivasilar interstitial opacities (General disorders) | 1 (1)
Hernia (Gastrointestinal disorders) | 1 (1)
Rotation of right foot (Musculoskeletal and connective tissue disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Complete hearing loss (Ear and labyrinth disorders) | 1 (1)
Ear infection (Ear and labyrinth disorders) | 1 (1)
Elevated alkaline phosphatase (Blood and lymphatic system disorders) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Facial numbness (Nervous system disorders) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Increased red blood cell distribution width (Blood and lymphatic system disorders) | 2 (2)
Elevated platelet count (Blood and lymphatic system disorders) | 2 (3)
Depression (Psychiatric disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Elevated Blood urea nitrogen (Blood and lymphatic system disorders) | 1 (2)
Hypocalcemia (Blood and lymphatic system disorders) | 2 (2)
Low hematocrit (Blood and lymphatic system disorders) | 2 (2)
Low erythrocytes (Blood and lymphatic system disorders) | 2 (2)
increased alanine aminotransferase (ALT) (Blood and lymphatic system disorders) | 2 (2)
Degenerative arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Ptosis, unilateral (Eye disorders) | 1 (1)
Cataract, unilateral (Eye disorders) | 1 (1)
Atypical urothelial cells in urine (Renal and urinary disorders) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Low Chloride (Blood and lymphatic system disorders) | 1 (1)
Clear cell cystic renal cell cancer (Renal and urinary disorders) | 1 (1)
Ehrlichiosis (Infections and infestations) | 1 (1)
Oral dysesthia (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study target enrollment was anticipated for 90 participants but only 23 participants completed treatment before study was terminated. The study was terminated due to insufficient resources and funding to support continuation of the trial. PI decision to terminate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT04398368/Prot_SAP_000.pdf